CLINICAL TRIAL: NCT06103539
Title: Pacertool-Study - Safety and Performance of the Presens-Catheter and the Pacer Software
Brief Title: Pacertool Early Feasibility Study - Safety and Performance
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pacertool AS (Industry)
Responsible Party: Sponsor
Other Study IDs: PaCRTool-Study 012023
Record Dates: First submitted 2023-10-23; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Dyssynchrony; Medical Device Performance
Keywords: Early feasibility observational study
MeSH Terms: interventions — Cardiac Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- 1: Patients with an indication for left heart catheterization or cardiac resynchornization therapy
  Interventions: Device: Cardiac catheterization and evoked response to cardiac stimulation

INTERVENTIONS:
Device: Cardiac catheterization and evoked response to cardiac stimulation — Cardiac catheterization with a combined elecrtophysiology and pressure sensing catheter to perform multisite stimulation and measure the evoked pressure response in a connected software.

SUMMARY:
The study is a non-randomized, two-part, open label, prospective single-site, single arm, safety and performance study. The study is designed to collect acute and long-term clinical data and user reported outcome data from using the PreSens-Catheter and PACER Software during cardiac catheterization and Cardiac Resynchronization Therapy (CRT) device implantation procedures. Subjects with indication for arterial catheterization and CRT will be included.

DETAILED DESCRIPTION:
The study consists of two parts:

1. Initial safety assessment: at least 5 patients undergoing coronary angiography or left heart catheterization and 5 patients undergoing cardiac resynchronization therapy device implantation to demonstrate acute safety and performance of the PreSens-Catheter and the PACER Software for Td measurements.
2. Safety and performance assessment: At least 35 patients with an indication for CRT implantation according to standard of care to demonstrate acute safety and performance of using the PreSens-Catheter and the PACER Software to measure Td and detect Synergy and Dyssynergy from multisite stimulation, and its utility to deliver measurements for the discrimination of two clinical cardiac reverse volumetric remodeling phenotypes based on Synergy and Dyssynergy in the targeted population.

Subjects will be followed for the duration of the procedure up to 24 hours for any serious adverse events, and subjects receiving a CRT device will be followed for 30 days follow-up for procedure or device-related events and for up to 6 months for cardiac volumetric remodeling phenotyping.

Clinical outcomes: Clinical outcome will be measured as Safety for the placement of the PreSens-Catheter, safety for the PreSens-Catheter and PACER Software combined for the measurement of Td and detection of Synergy/ Dyssynergy from stimulation, and diagnostic/ predictive performance of the PreSens-Catheter and PACER Software with the measurement of end-systolic volume at 6-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

Part I:

* Subject has an indication for coronary angiography or left heart catheterization or cardiac resynchronization therapy.
* QRS duration between 90-150ms.
* Subject is ≥ 18 years old.
* Willingness, ability, and commitment to participate in baseline and follow-up evaluations for the full duration of the clinical study.
* Willing and able to give informed consent.

Part II:

* Subject in sinus rhythm with an indication for implantation of a Cardiac Resynchronization Device (Appendix I)
* NYHA Class II-IV (Ambulatory IV)
* EF<35%
* QRS duration >120ms.
* Subject is ≥ 18 years old.
* Willingness, ability, and commitment to participate in baseline and follow-up evaluations for the full duration of the clinical study.
* Willing and able to give informed consent.

Exclusion Criteria:¨

* Subject has unstable angina/ acute coronary ischemia/ infarction
* Previous myocardial infraction (<6 months)
* History of blood clothing or bleeding disease
* Prior history of documented cerebral infarction, TIA or systemic embolism (excluding a postoperative DVT)
* Subject has an arterial unstable aneurysm
* Subject has severe peripheral vascular disease
* Subject has an artificial aortic or mitral valve replacement
* Subject has severe aortic valve disease
* Subject has a clinically significant infection (bacteriemia or sepsis)
* Subject has contraindications to anticoagulation
* Patients with a serious allergy to drugs necessary for the procedure such as anticoagulants and protamine
* Subject has left atrial/ ventricular thrombus
* Patients with severe vascular obstructions in the desired/ presumed insertion path of the catheter
* Significant or symptomatic hypotension
* NYHA class IV (hospitalized), severe circulation instability or shock
* Ongoing/ persistent atrial arrythmias
* History of Rheumatic fever
* Subject has sensitivity to contrast media
* Contraindications to CT or fluoroscopy
* Distorted cardiac anatomy due to congenital heart disease
* Pregnant or possibly pregnant
* Not eligible for thoracotomy procedures
* Life expectancy <1 years
* Any other condition that, in the judgement of the investigator, makes the subject a poor candidate for this procedure, the study or compliance with the protocol (includes addictive disease, extensive travel away from the research center)
* Clinically significant psychological condition that in the investigator's opinion would prohibit the subject's ability to meet the protocol requirements
* Current enrollment in any other study protocol where testing or results from that study may interfere with the procedure or outcome measurements of this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is adult patients (>18years) with (part I) an indication for left heart catheterization, or (part I and II) a clinical syndrome of heart failure with reduced ejection fraction and normal sinus rhythm with signs of ventricular electrical conduction defects in the heart, who meets standard criteria for implantation of a cardiac resynchronization therapy device.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Outcome (PreSens-Catheter): | 24 hours
  The primary safety outcome is the incidence of procedure or device-related Serious Adverse Events (SAEs and SADEs) on the day of the procedure
Primary Safety Outcome Measures (PreSens-Catheter and PACER Software): | 4 hours
  The primary safety outcome of the PreSens-Catheter and PACER Software is the incidence of false positive readings of Synergy resulting from multisite stimulation from PreSens-Catheter in patients with narrow QRS and false negative readings (Dyssynergy) compared to the resulting reading from pacing with the CRT device.
Primary Performance Outcome Measures (PreSens-Catheter and PACER Software): | 6 months
  Detection of Synergy and Dyssynergy to phenotype patients for the prediction of reverse volumetric remodeling response after 6 months of Cardiac Resynchronization Therapy. Outcome is based on the change in End-Systolic Volume (ESV) from baseline to 6 months follow-up in the respective phenotypes. The study is powered to detect a ΔESV of 30% points difference between the Synergy and Dyssynergy characterized patients after 6 months of Cardiac Resynchronization Therapy.

SECONDARY OUTCOMES:
Safety Outcome Measures (PreSens-Catheter): | 30 days
  Percentage of subjects experiencing a composite safety event. The composite safety outcome (CSO) defined as the incidence of events which are device- or procedure-related
Performance Outcome Measures (PreSens-Catheter) | 4 hours
  a) The proportion of subjects that achieve Acute Procedural Success (APS) defined as the correct insertion and placement of the PreSens-Catheter within the heart with confirmed readings/ recordings from the catheter and imaged with fluoroscopy in two planes, in at least one of the defined positions depending on available access sheets (on an intention-to-treat basis). b) The proportion of subjects that had the PreSens-Catheter placed in the left heart with the intention to place the catheter with the distal electrodes in three different positions (anterior, lateral, posterior); number of positions achieved in each patient. c) Product performance evaluated on a 5-point semi-quantitative scale ("strongly disagree" to "strongly agree") [Time Frame: During Procedure]. d) Acute product performance will be quantitatively and qualitatively evaluated during the procedure.
Performance Outcome Measures (PreSens-Catheter and PACER Software): | 4 hours
  The proportion of subjects that achieve Acute Procedural Success (APS) defined as successful placement of the PreSens-Catheter in the heart and measurement of Td (time to peak exponential pressure rise (dP/dt)) with the PACER Software; with stimulation from the PreSens-Catheter and from the CRT (with the rate of agreement) with the PreSens-Catheter placed in at least two out of three defined positions. (CRT recipients only).

OTHER OUTCOMES:
iv) Exploratory Performance Outcome Measures (PreSens-Catheter and PACER Software): | 4 hours
  (a) Percentage of subjects experiencing (from each position in the left heart): (i) Demonstration of prolongation of Td with pacing off a proximal electrode (ii) Demonstration of prolongation of Td with pacing off a distal electrode (iii) Demonstration of shortening of Td (Synergy) with pacing from electrodes from both electrode groups (distal and proximal) compared to the shortest Td with pacing from either distal or proximal electrode. (iv) Demonstration of shortening of Td (Synergy) with pacing from electrodes from both electrode groups (distal and proximal) compared to baseline Td in patients with QRS duration above 130ms and below or equal to 130ms. (v) Demonstration of prolongation of Td (Dyssynergy) with biventricular pacing (negative responder, true negative result) compared to baseline Td in patients with QRS duration above 130ms and ≤130ms. (vi) Demonstration of a short Td (≤120ms) at baseline in patients with a QRS duration ≤130ms and long Td (>120ms) at baseline in patient

CONTACTS AND LOCATIONS:
Overall Officials: Tamaz Shaburishvili, MD, Principal Investigator — Tbilisi Heart and Vascular Clinic
Locations (1):
- Tbilisi Heart and Vascular Clinic, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Odland HH, Holm T, Cornelussen R, Kongsgard E. Determinants of the time-to-peak left ventricular dP/dt (Td) and QRS duration with different fusion strategies in cardiac resynchronization therapy. Front Cardiovasc Med. 2022 Sep 15;9:979581. doi: 10.3389/fcvm.2022.979581. eCollection 2022. PMID 36186985
- [Background] Odland HH, Villegas-Martinez M, Ross S, Holm T, Cornelussen R, Remme EW, Kongsgard E. Shortening of time-to-peak left ventricular pressure rise (Td) in cardiac resynchronization therapy. ESC Heart Fail. 2021 Dec;8(6):5222-5236. doi: 10.1002/ehf2.13601. Epub 2021 Sep 12. PMID 34514746